CLINICAL TRIAL: NCT01043393
Title: An Open Label, Safety/Efficacy Study to Assess the Potential for Adrenal Suppression Following Multiple Dosing With Desoximetasone 0.25% Topical Spray in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Desoximetasone Spray 0.25%, Hypothalamic Pituitary Adrenal (HPA) Axis Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSXS-0805; Study # 70915005 (Other: Novum)
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Psoriasis
Keywords: Plaque psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Desoximetasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psoriasis involving 10-15% BSA (Experimental): Patients 18 years of age or older with a confirmed diagnosis of moderate to severe plaque psoriasis having involvement of 10-15% of their body surface area.
  Interventions: Drug: Desoximetasone 0.25% spray
- Psoriasis involving >15% of BSA (Experimental): Patients 18 years of age or older with a confirmed diagnosis of moderate to severe plaque psoriasis having involvement of >15% of their body surface area.
  Interventions: Drug: Desoximetasone 0.25% spray

INTERVENTIONS:
Drug: Desoximetasone 0.25% spray — Desoximetasone spray applied to affected areas twice daily for 28 days

SUMMARY:
The objective of this study is to evaluate the potential of desoximetasone 0.25% topical spray to suppress HPA axis function. The potential for adrenal suppression will be assessed following multiple dosing with Desoximetasone 0.25% Topical Spray in patients with moderate to severe plaque psoriasis. The secondary objectives are to evaluate the efficacy parameters and to evaluate the adverse event (AE) profile.

ELIGIBILITY:
Inclusion Criteria:

* Have a definite clinical diagnosis of stable plaque psoriasis with the extent of BSA affected as designated for each group
* Group 1: involvement of 10-15% of their BSA
* Group 2: involvement of > 15% of their BSA
* Have a Physicians Global Assessment (PGA) score of 3 (moderate) or 4 (severe) at baseline for the overall disease severity.
* Results from a cortisol response test that are considered normal and show no evidence of any abnormal HPA function or adrenal response. Patients must fulfill all of these stipulations:

Exclusion Criteria:

* Female who is pregnant, nursing, planning to become pregnant during the duration of the study, or if of child bearing potential and sexually active not prepared to use appropriate contraceptive methods to avoid pregnancy.
* Patient has current diagnosis of types of psoriasis other than stable plaque psoriasis (i.e. acute, guttate, erythrodermic, exfoliative or pustular psoriasis) or has psoriasis of any kind on the face or scalp that will require active treatment during the study.
* Patient has a history of psoriasis that has been unresponsive to topical corticosteroid therapy.
* In the Investigator's opinion, the patient has other dermatological conditions, such as atopic or contact dermatitis, that may interfere with the clinical assessments of the signs and symptoms of psoriasis
* Patient has a history of allergy or sensitivity to corticosteroids or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the patient or the results of the study.
* Patient has a history of an adverse reaction to CortrosynTM or similar test reagents.
* Patient has a significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participation in the study.
* Patient is currently receiving or has received any radiation therapy, anti-neoplastic agents or immunosuppressant medication within 4 weeks prior to the first dose of study drug.
* Patient has undergone treatment with any systemic or photo antipsoriatic therapy within 8 weeks of the first dose of study drug.
* Patient has been treated within 12 weeks (or five half lives whichever is less) prior to the first dose of study drug with any biological therapies for psoriasis.
* Patient has received any systemic steroids within 4 weeks of the first dose of the study drug.
* Patients who have used any topical antipsoriatic agents of any kind or any topical corticosteroids for any reason within 2 weeks prior to first use of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Investigator Site, Hot Springs, Arkansas
  - Investigator Site, Albuquerque, New Mexico
  - Investigator Site, Simpsonville, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Psoriasis Involving 10-15% BSA: Patients 18 years of age or older with a confirmed diagnosis of moderate to severe plaque psoriasis having involvement of 10-15% of their body surface area (BSA).
  Desoximetasone 0.25% spray: Desoximetasone spray applied to affected areas twice daily for 28 days
- Psoriasis Involving >15% of BSA: Patients 18 years of age or older with a confirmed diagnosis of moderate to severe plaque psoriasis having involvement of >15% of their body surface area (BSA).
  Desoximetasone 0.25% spray: Desoximetasone spray applied to affected areas twice daily for 28 days
Period: Overall Study
Arm/Group | Psoriasis Involving 10-15% BSA | Psoriasis Involving >15% of BSA
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psoriasis Involving 10-15% BSA | Psoriasis Involving >15% of BSA | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Median (Full Range); unit: years] | 52.08 (3.55) [18 to 74] | 46.75 (5.99) [18 to 74] | 49.42 (4.77) [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients in the Study With Hypothalamic Pituitary Adrenal (HPA) Axis Suppression
Description: Each patient is assessed at Day 28. A cortisol response test performed at baseline are reevaluated at the conclusion of the study. If the normal cortisol response test measured at baseline is no long present the patient is considered to have demonstrated possible HPA axis suppression.
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Psoriasis Involving 10-15% BSA | Psoriasis Involving >15% of BSA
Number analyzed (Participants) | 12 | 12
participants | 2 (3.55) | 3 (5.99)
Statistical Analysis 1: Comparison: Psoriasis Involving 10-15% BSA vs Psoriasis Involving >15% of BSA; Test type: Superiority or Other; Odds Ratio (OR) = 0.779, 95% CI 2-sided [0.055 to 11.126]

2. Secondary Outcome: Change From Baseline in Percent Body Surface Area (%BSA) Affected by Psoriasis
Description: Body Surface Area (BSA) is a numerical score used to measure the physician's assessment of the percentage of the participant's total BSA involved with psoriasis.
  BSA = SQRT ((height (cm) X weight (kg))/3600)
  BSA is in m2, W is weight in kg, and H is height in cm. Total body Surface Area (BSA) in meters squared
  %Body Surface Area Affected the "Rule of Nine" was be used
Time Frame: 28 days
Population: No statistical analysis provided for Percentage of Body Surface Area Affected by Psoriasis.
  As the study is not powered sufficiently to perform efficacy statistical analysis, descriptive statistical analysis are presented on the mean change from baseline in % BSA affected
Measure: Mean (Standard Deviation); unit: percentage of Body Surface Area Affected
Arm/Group | Psoriasis Involving 10-15% BSA | Psoriasis Involving >15% of BSA
Number analyzed (Participants) | 12 | 12
percentage of Body Surface Area Affected | 5.50 (3.55) [0.0338 to 11.126] | 3.50 (5.99) [0.0921 to 1.168]

3. Secondary Outcome: Change From Baseline in Physician's Global Assessment (PGA) Score for Psoriasis
Description: The PGA scale is designed to evaluate the physician's global assessment of the participant's psoriasis based on severity of induration,erythema and scaling. The PGA is assessed on a scale of 0 to 5 (0 = clear, 5 = severe).
Time Frame: 28 days
Population: No statistical analysis provided for Percentage of Participants With a Physician's Global Assessment (PGA) of Psoriasis Score of 0 (Clear) or 1 (Almost Clear)
Measure: Mean (Standard Deviation); unit: percentage of physician's global assessm
Arm/Group | Psoriasis Involving 10-15% BSA | Psoriasis Involving >15% of BSA
Number analyzed (Participants) | 12 | 12
percentage of physician's global assessm | 1.83 (0.94) | 1.33 (1.15)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Psoriasis Involving 10-15% BSA | Psoriasis Involving >15% of BSA
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psoriasis Involving 10-15% BSA (N=12) | Psoriasis Involving >15% of BSA (N=12)
Adrenal Suppression (Endocrine disorders) | 2 (2) | 3 (3)
Application Site Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sciatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No